CLINICAL TRIAL: NCT01276353
Title: A Randomized, Double Blind, Parallel-Group Comparison Study Versus E2020 10mg Followed by an Open-label Extension Phase to Explore the Safety of E2020 SR 23 mg in Japanese Subjects With Severe Alzheimer's Type Dementia
Brief Title: A Study Versus E2020 10mg Followed by an Open-label Extension Phase to Explore the Safety of E2020 SR 23 mg in Japanese Subjects With Severe Alzheimer's Type Dementia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: E2020-J081-221
Record Dates: First submitted 2011-01-12; First posted 2011-01-13 (Estimated); Results first posted 2014-08-01 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2014-08

CONDITIONS: Alzheimer's Type Dementia
Keywords: Alzheimer Disease; Dementia; Delirium; Amnestic; Cognitive Disorders; Donepezil; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Tauopathies; Neurodegenerative Diseases; Mental Disorders; Cholinesterase Inhibitors; Enzy
MeSH Terms: conditions — Alzheimer Disease; Dementia; Delirium; Cognitive Dysfunction; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Tauopathies; Neurodegenerative Diseases; Mental Disorders | interventions — Donepezil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: E2020
- 2 (Active Comparator)
  Interventions: Drug: E2020

INTERVENTIONS:
Drug: E2020 — Patients will take study medication orally, once daily, for 2 weeks according to a double-dummy design in the double blind phase: 23 mg donepezil sustained release (SR) concurrently with placebo identical in appearance to the 10 mg donepezil immediate release (IR) formulation
  Arms: 1
Drug: E2020 — 10 mg donepezil immediate release (IR) concurrently with placebo identical in appearance to the 23 mg donepezil sustained release (SR) formulation. All patients who complete the double blind phase will take 23 mg donepezil sustained release (SR) orally, once daily, for 52 weeks in the Open-label Extension phase.
  Arms: 2

SUMMARY:
The purpose of this study is to compare 23 mg donepezil sustained release (SR) to the currently marketed formulation of 10 mg donepezil immediate release (IR) in patients with severe Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria

* Diagnostic evidence of probable Alzheimer's disease (AD) consistent with the Diagnostic and Statistical Manual for Mental Disorders-version IV (DSM-IV)
* Hachinski Ischemic Score
* Functional Assessment Staging (FAST) scale greater than or equal to 6 at Screening.
* Mini-Mental State Examination (MMSE) score of 1 to 12 at Screening
* Subjects who are on a stable Aricept- dose of 10 mg immediate release (IR), taken as a single, daily dose for 3 months prior to the Screening Visit
* Evidence consistent with Alzheimer's disease (AD) on any cranial image on magnetic resonance imaging (MRI) or computed tomography (CT) scan or etc. obtained within 24 months prior to the Screening Visit. Subjects who have any observations of dementia other than Alzheimer's type after the last image diagnosis should be reconfirmed.
* Age 50 years
* Written informed consent is to have been obtained from the subject (if possible) or from the subject's legal guardian or other representative

Exclusion Criteria

* Subjects with dementia other than Alzheimer's type
* Subjects with significant neurological or psychiatric disorders such as stroke, brain tumor, schizophrenia, epilepsy, normal pressure hydrocephalus, mental retardation, a history of head injury with loss of consciousness, or a history of brain surgery followed by persistent deficits
* Subjects with allergy to donepezil hydrochloride or piperidine derivatives
* Subjects with a cause of Alzheimer's disease (AD) which is supported by any laboratory tests such as Vitamin B12, folate levels, triiodothyronine, free triiodothyronine, thyroxine, thyroid stimulating hormone (TSH) or serologic test for syphilis

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2011-01; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naoki Kubota, Study Director — Neuroscience Clinical Development Section. JAC PCU. Eisai Co., Ltd.
Locations (11):
- Japan (11):
  - Akita, Akita
  - Fukuoka, Fukuoka
  - Kitakyushu, Fukuoka
  - Mizunami, Gifu
  - Yokosuka, Kanagawa
  - Sanjō, Niigata
  - Kurashiki, Okayama-ken
  - Saitama, Saitama
  - Fuji, Shizuoka
  - Hachiōji, Tokyo
  - Kodaira, Tokyo

RESULTS

PARTICIPANT FLOW:
Groups:
- E2020 SR 23 mg: E2020 SR 23 mg 1 tablet + E2020 10 mg placebo tablet once daily in the morning for 2 weeks in the double-blind phase. E2020 SR 23 mg once daily in the morning for 52 weeks in the extension phase.
- E2020 10 mg: E2020 10 mg 1 tablet + E2020 SR 23 mg placebo tablet once daily in the morning for 2 weeks in the double-blind phase. E2020 SR 23 mg once daily in the morning for 52 weeks in the extension phase.
Period: Double-blind
Arm/Group | E2020 SR 23 mg | E2020 10 mg
Started | 22 | 23
Completed | 19 | 23
Not Completed | 3 | 0
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Extension
Arm/Group | E2020 SR 23 mg | E2020 10 mg
Started | 19 | 23
Completed | 12 | 14
Not Completed | 7 | 9
Not completed — Adverse Event | 2 | 5
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Withdrawal of study drug 4 days in a row | 3 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Prohibited concomitant medications | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | E2020 SR 23 mg | E2020 10 mg | Total
Number analyzed (Participants) | 22 | 23 | 45
Age, Continuous [Mean (Standard Deviation); unit: Years] | 79.3 (9.8) | 73.6 (10.8) | 76.4 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 32
  Male | 6 | 7 | 13
Hachinski Score [Mean (Standard Deviation); unit: Scores on a Scale] — The Hachinski Ischaemic Score (HIS) is an attempt to differentiate Alzheimer's type dementia and multi-infarct dementia. It uses a system of 13 features of with a score of 1 or 2, adding the scores together for a final score. A cut-off score less than or equal to 4 for Dementia of Alzheimer's Type (DAT) and greater than or equal to 7 for Vascular Dememntia (VaD) has a sensitivity of 89% and a specificity of 89%.
  Scores on a Scale | 1.1 (1.3) | 0.7 (1.1) | 0.9 (1.2)

OUTCOME MEASURES:

1. Secondary Outcome: Cmax of E2020 on Visits 2 and 3 According to Cytochrome P450 2D6 (CYP2D6) Phenotype Status
Description: All subjects were identified as Extensive Metabolizer [EM] or Intermediate Metabolizer [IM] predicted from their CYP2D6 phenotypes. Ultra-rapid Metabolizer (UM) and Poor Metabolizer (PM) were not identified in any subject. Since the analysis population i
Time Frame: Visit 2 [Day1] and Visit 3 [Day 15]
Population: Pharmacokinetic Analysis Set
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- E2020 10 mg (EM): E2020 10 mg 1 tablet + E2020 SR 23 mg placebo tablet once daily in the morning for 2 weeks in the double-blind phase. E2020 SR 23 mg once daily in the morning for 52 weeks in the extension phase.
Arm/Group | E2020 SR 23 mg | E2020 10 mg (EM)
Number analyzed (Participants) | 22 | 23
ng/mL
  Visit 2 EM [IR: n=16, SR: n=17] | 117.999 (28.898) | 98.117 (32.323)
  Visit 2 IM [IR: n=5, SR: n=4] | 161.363 (18.761) | 104.294 (23.962)
  Visit 3 EM [IR: n=16, SR: n=15] | 116.771 (31.663) | 63.896 (20.662)
  Visit 2 IM [IR: n=5, SR: n=3] | 182.953 (48.422) | 79.802 (24.984)

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of E2020 on Visits 2 and 3
Time Frame: Visit 2 [Day1] and Visit 3 [Day 15]
Population: Pharmacokinetic Analysis Set: the group of subjects who had received at least one quantifiable E2020 concentration in plasma
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- E2020 SR 23 mg: E2020 SR 23 mg 1 tablet + E2020 10 mg placebo tablet once daily in the morning for 2 weeks in the double-blind phase. E2020 SR 23 mg once in the morning daily for 52 weeks in the extension phase.
Arm/Group | E2020 SR 23 mg | E2020 10 mg
Number analyzed (Participants) | 22 | 23
ng/mL
  Visit 2 | 126.503 (31.27) | 97.006 (32.934)
  Visit 3 | 127.335 (40.654) | 66.081 (24)

ADVERSE EVENTS:
Time Frame: Up to 54 weeks
Groups:
- E2020 SR 23 mg (Double-blind): E2020 SR 23 mg 1 tablet + E2020 10 mg placebo tablet once daily in the morning for 2 weeks in the double-blind phase.
- E2020 10 mg (Double-blind): E2020 10 mg 1 tablet + E2020 SR 23 mg placebo tablet once daily in the morning for 2 weeks in the double-blind phase.
- E2020 SR 23 mg (Extension); E2020 10 mg (Extension): E2020 SR 23 mg once daily in the morning for 52 weeks in the extension phase.
Arm/Group | E2020 SR 23 mg (Double-blind) | E2020 10 mg (Double-blind) | E2020 SR 23 mg (Extension) | E2020 10 mg (Extension)
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/23 | 0/19 | 1/23
Other Adverse Events (participants affected / at risk) | 13/22 | 2/23 | 9/19 | 16/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | E2020 SR 23 mg (Double-blind) (N=22) | E2020 10 mg (Double-blind) (N=23) | E2020 SR 23 mg (Extension) (N=19) | E2020 10 mg (Extension) (N=23)
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | E2020 SR 23 mg (Double-blind) (N=22) | E2020 10 mg (Double-blind) (N=23) | E2020 SR 23 mg (Extension) (N=19) | E2020 10 mg (Extension) (N=23)
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 2 | 0
Nausea (Gastrointestinal disorders) | 3 | 1 | 0 | 7
Vomiting (Gastrointestinal disorders) | 4 | 1 | 0 | 7
Electrocardiogram QT prolonged (Investigations) | 2 | 0 | 1 | 0
Weight decreased (Investigations) | 2 | 0 | 3 | 1
Decreased appetite (Metabolism and nutrition disorders) | 6 | 0 | 3 | 4
Somnolence (Nervous system disorders) | 2 | 0 | 1 | 4
Eye Discharge (Eye disorders) | 0 | 0 | 1 | 0
Epulis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Oedema (General disorders) | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0
Blood pressure decreased (Investigations) | 0 | 0 | 1 | 0
Blood pressure increased (Investigations) | 0 | 0 | 1 | 0
Blood uric acid increased (Investigations) | 1 | 0 | 1 | 0
Dyskinesia (Nervous system disorders) | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other